CLINICAL TRIAL: NCT00893672
Title: A Cluster-Randomized Two-Period Cross-Over Study Comparing Routine and on-Demand Prescription of Chest Radiographs in Mechanically Ventilated Adults : the RARE Study
Brief Title: Comparison of Two Chest Radiograph Prescription Strategies in Intensive Care Unit
Acronym: RARE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Zakia IDIR, Department Clinical Research of Developpement
Other Study IDs: SCR06006
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Last update posted 2009-05-06 (Estimated); Status verified 2009-05

CONDITIONS: Patient Care; Quality of Health Care; Intensive Care Units; Ventilation, Mechanical
Keywords: Radiography, Thoracic; Intensive Care Units; Ventilation, mechanical; Matched-Pair Analysis
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Routine strategy of chest radiograph prescription
- 2: On-demand strategy of chest radiograph prescription

SUMMARY:
Current guidelines recommend Routine daily chest radiographs (CXRs) for mechanically ventilated patients in intensive care units (ICUs). However, some ICUs have shifted to an On-demand strategy, in which this CXR is only prescribed if warranted by the patient's status at the morning physical examination. Here the investigators compared Routine and On-demand strategies in 21 French ICUs. The working hypothesis was that CXR prescriptions would fall by at least 20% with the On-demand strategy, with no reduction in quality of care.

DETAILED DESCRIPTION:
Based on a cluster-randomized two-period two-strategies cross-over design, respectively 11 and 10 participating ICUs applied the Routine and On-demand strategies during the first period, each enrolling 20 consecutive patients requiring mechanical ventilation for at least two days. Each ICUs applied then applied the alternative strategy during the second period, again enrolling 20 consecutive patients.

ELIGIBILITY:
Inclusion Criteria:

* All newly admitted adult patients receiving mechanical ventilation at the time of the morning visit-any day during their ICU stay

Exclusion Criteria:

* Patients with mechanical ventilation lasting less than 2 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All newly admitted adult patients receiving mechanical ventilation at the time of the morning visit in ICU
Sampling Method: Probability Sample
Enrollment: 849 (Actual)
Dates: Start 2006-12; Primary Completion 2007-08 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Average number of chest radiographs per patient-day during mechanical ventilation | Every patient-day during mechanical ventilation.

SECONDARY OUTCOMES:
Mortality rate in ICU | During the inpatient stay in ICU
Average length of stay | During the inpatient stay in ICU
Average duration of mechanical ventilation | During the inpatient stay in ICU
Number of radiographs with new findings leading to therapeutic or diagnostic interventions | During the inpatient stay in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand GUIDET, MD PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Saint-Antoine, Paris, Paris, France

REFERENCES:
- [Derived] Hejblum G, Chalumeau-Lemoine L, Ioos V, Boelle PY, Salomon L, Simon T, Vibert JF, Guidet B. Comparison of routine and on-demand prescription of chest radiographs in mechanically ventilated adults: a multicentre, cluster-randomised, two-period crossover study. Lancet. 2009 Nov 14;374(9702):1687-93. doi: 10.1016/S0140-6736(09)61459-8. Epub 2009 Nov 4. PMID 19896184